CLINICAL TRIAL: NCT06283446
Title: Enhancing Prospective Thinking in Early Recovery
Brief Title: Enhancing Prospective Thinking in Early Recovery (NERF)
Acronym: NERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Brandon G. Oberlin, PhD, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1805574553; Aims 11-13; 1R21AA029760-01 (NIH)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Masking Description: Eligible participants will be randomly assigned to either the high-intensity (experimental) or low-intensity (control) groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity (Experimental): Participants will receive high-intensity episodic future-thinking cue images, and high-intensity episodic recent-thinking cue images during an MRI decision-making task.
  Interventions: Behavioral: High-Intensity Cue
- Low-Intensity (Control) (Active Comparator): Participants will receive low-intensity episodic future-thinking cue images, and low-intensity episodic recent-thinking cue images during an MRI decision-making task.
  Interventions: Behavioral: Low-Intensity Cue

INTERVENTIONS:
Behavioral: High-Intensity Cue — Participants in the high-intensity group will receive high-intensity image cues that represent self-reported events they did on the previous day and self-reported events they look forward to in the future.
  Arms: High-Intensity
Behavioral: Low-Intensity Cue — Participants in the low-intensity group will receive low-intensity image cues that represent self-reported events they did on the previous day and self-reported events they look forward to in the future.
  Arms: Low-Intensity (Control)

SUMMARY:
The goal of this clinical trial is to test the prosocial effects of personally-relevant, high-intensity episodic future-thinking (EFT) cues in alcohol use disorder persons and related brain mechanisms. The main question[s] this trial aims to answer are:

Will high-intensity EFT cues will produce greater delayed reward preference than low-intensity cues? Will high-intensity EFT cues effect greater treatment-seeking interest? Will high-intensity EFT cues elicit greater response in regions for prospective thinking during delay discounting (vs. low-intensity) Will nucleus accumbens-precuneus resting connectivity correlate with behavioral SS? Will the novel behavioral SS decision-making task activate the nucleus accumbens? Researchers will compare the experimental (high-intensity group) and control (low-intensity) groups to see if there are differences in the results for the questions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Abstinence between 30 days ≤ 1 year
* Verbal endorsement of commitment to recovery
* English comprehension

Exclusion Criteria:

* Unstable medical disorders
* Outside the age range of 18-60
* Habitual substance or alcohol use
* Smell/taste disorders
* Unstable psychiatric conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Increase Prospective Thinking | [Time Frame: Study Day Visit (Day 1)]
  High-intensity episodic future-thinking image cues will increase prospective thinking.
Delayed Rewards | [Time Frame: Study Day Visit (Day 1)]
  High-intensity episodic future-thinking image cues will change preference for delayed rewards, which will be measured using a behavioral delayed discounting task.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Oberlin, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine - Goodman Hall, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared in accordance with the National Institutes of Health National Data Archive requirements and upon the consent of the study participant.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared at the specified submission deadlines assigned by the National Institutes of Health (typically every April or October). Data will be available upon the discretion of the National Institutes of Health.
Access Criteria: No individually identifiable participant data will be submitted to the National Data Archive. All collected participant data is de-identified, and will be made available for other researchers to use upon requests submitted through the National Data Archive portal, and approval from the principal investigator.